CLINICAL TRIAL: NCT00913978
Title: A Prospective Randomized Evaluation of Two Perioperative Active Warming Techniques in Maintenance of Normothermia in Colorectal Surgeries
Brief Title: Perioperative Active Warming Techniques in Colorectal Surgeries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to financial status of sponsor.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Meltem Yilmaz, Associate Professor in Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00202644
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Normothermia
Keywords: Normothermia; Colorectal Surgery; Bair Huggers; VitaHeat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1: VitaHeat (Active Comparator): Patients in group one will be warmed perioperatively with the VitaHeat mattress and IV fluid warmers once they are in the operating room.
  Interventions: Device: Group 1: VitaHeat
- Group 2: Bair Hugger (Active Comparator): Patients in group two will be warmed perioperatively with the upper body bair hugger and IV fluid warmers once they are in the operating room.
  Interventions: Device: Group 2: Bair Hugger

INTERVENTIONS:
Device: Group 1: VitaHeat — Patients will receive active warming via a heating mattress (VitaHEAT Medical) placed on the OR table with two thin sheets between the patient and the device; one covering the mattress and the other used as the draw sheet as usual practice. The device will be turned on 10 minutes prior to the patients' arrival to the operating room table. Patients' upper body will be covered with blankets. To increase skin surface contact with the mattress any blankets remaining under the patients' chest or head will be removed after intubation and replaced with a donut. IV fluid warmer initiated on arrival to the operating room. The operating room temperatures will be adjusted to 21°C.
  Arms: Group 1: VitaHeat
Device: Group 2: Bair Hugger — Patients will receive standard forced air warming applied to the upper body and turned on after the patient is prepped and draped. These warmers will be placed directly in contact with the skin without any intervening insulation. IV fluid warmer initiated on arrival to the operating room. The operating room temperatures will be adjusted to 21°C.
  Arms: Group 2: Bair Hugger

SUMMARY:
We propose a study in which we compare two intraoperative active warming devices for maintenance of normothermia in patients undergoing colorectal surgery. A novel underbody resistive warming mattress (VitaHeat) will be compared to the forced air warming blanket (3M Bair Hugger) that is currently used in our institution. Our hypothesis is that the underbody resistive warming mattress will be equally effective as forced air warming in maintaining normothermia in colorectal surgery.

DETAILED DESCRIPTION:
Stratified randomization will be performed using a computerized randomization table where the strata will be type of surgery (open vs closed) and the treatment will be forced air blanket or underbody mattress warming device. This will allow equal groups of both warming devices in both types of surgery.

Group 1: Patients will receive active warming via a heating mattress (VitaHEAT Medical) placed on the OR table with two thin sheets between the patient and the device; one covering the mattress and the other used as the draw sheet as usual practice. The device will be turned on 10 minutes prior to the patients' arrival to the operating room table. Patients' upper body will be covered with blankets. To increase skin surface contact with the mattress any blankets remaining under the patients' chest or head will be removed after intubation and replaced with a donut.

Group 2: Patients will receive standard forced air warming applied to the upper body and turned on after the patient is prepped and draped. These warmers will be placed directly in contact with the skin without any intervening insulation.

Both groups will have IV fluid warmer initiated on arrival to the operating room. The operating room temperatures will be adjusted to 21°C.

Participation in the study is voluntary. The patients may choose not to enroll in the research. Patients who choose not to enroll will use the standard forced air warmer.

Preoperative and postoperative temperatures will be measured orally. Intraoperative core and skin temperatures will be monitored continuously at 1 minute intervals using an esophageal probe and skin temperature probe using a skin temp probe placed on the great toe and covered to prevent any contact with the warming devices.

Intraoperative period: The participants temperature will be monitored and documented at prescribed times.

Postoperative period: The participants will have temperature monitored in the post anesthesia care area.

Participation in this study will last for 30 days following surgery at which point study member will call patient for a 2-4 minute phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old undergoing laparoscopic or open colorectal surgical procedures under general anesthesia.

Exclusion Criteria:

* Any patient who is less than 18 years old.
* Emergent surgery
* Any patient with thyroid problems
* Any patient with preoperative fever
* Any patient who is pregnant
* Any adult patients unable to consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meltim Yilmaz, M.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Torossian A. Thermal management during anaesthesia and thermoregulation standards for the prevention of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):659-68. doi: 10.1016/j.bpa.2008.07.006. PMID 19137809
- [Background] Sessler DI, Schroeder M. Heat loss in humans covered with cotton hospital blankets. Anesth Analg. 1993 Jul;77(1):73-7. doi: 10.1213/00000539-199307000-00014. PMID 8317751
- [Background] Cheney FW, Posner KL, Caplan RA, Gild WM. Burns from warming devices in anesthesia. A closed claims analysis. Anesthesiology. 1994 Apr;80(4):806-10. doi: 10.1097/00000542-199404000-00012. PMID 8024134
- [Background] Taguchi A, Ratnaraj J, Kabon B, Sharma N, Lenhardt R, Sessler DI, Kurz A. Effects of a circulating-water garment and forced-air warming on body heat content and core temperature. Anesthesiology. 2004 May;100(5):1058-64. doi: 10.1097/00000542-200405000-00005. PMID 15114200
- [Background] Janicki PK, Higgins MS, Janssen J, Johnson RF, Beattie C. Comparison of two different temperature maintenance strategies during open abdominal surgery: upper body forced-air warming versus whole body water garment. Anesthesiology. 2001 Oct;95(4):868-74. doi: 10.1097/00000542-200110000-00014. PMID 11605926
- [Background] Hynson JM, Sessler DI. Intraoperative warming therapies: a comparison of three devices. J Clin Anesth. 1992 May-Jun;4(3):194-9. doi: 10.1016/0952-8180(92)90064-8. PMID 1610573
- [Background] Brauer A, Weyland W, Kazmaier S, Trostdorf U, Textor Z, Hellige G, Braun U. Efficacy of postoperative rewarming after cardiac surgery. Ann Thorac Cardiovasc Surg. 2004 Jun;10(3):171-7. PMID 15312013
- [Background] Smith CE, Desai R, Glorioso V, Cooper A, Pinchak AC, Hagen KF. Preventing hypothermia: convective and intravenous fluid warming versus convective warming alone. J Clin Anesth. 1998 Aug;10(5):380-5. doi: 10.1016/s0952-8180(98)00049-x. PMID 9702617
- [Background] Negishi C, Hasegawa K, Mukai S, Nakagawa F, Ozaki M, Sessler DI. Resistive-heating and forced-air warming are comparably effective. Anesth Analg. 2003 Jun;96(6):1683-1687. doi: 10.1213/01.ANE.0000062770.73862.B7. PMID 12760996
- [Background] Melton GB, Vogel JD, Swenson BR, Remzi FH, Rothenberger DA, Wick EC. Continuous intraoperative temperature measurement and surgical site infection risk: analysis of anesthesia information system data in 1008 colorectal procedures. Ann Surg. 2013 Oct;258(4):606-12; discussion 612-3. doi: 10.1097/SLA.0b013e3182a4ec0f. PMID 23989047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients were consented to participate, 4 were withdrawn from the study to leave an analysis sample of 46 subjects. The study was terminated early due to financial constraints from the sponsor.
Period: Overall Study
Arm/Group | Group 1: VitaHeat | Group 2: Bair Hugger
Started | 26 | 24
Completed | 25 | 21
Not Completed | 1 | 3
Not completed — Surgeon choice | 1 | 3

BASELINE CHARACTERISTICS:
Population: 1 subjects in the Vitaheat group and 3 subjects in the Bair Hugger group were not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: VitaHeat | Group 2: Bair Hugger | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Continuous [Mean (Full Range); unit: Years] | 58.36 [24 to 78] | 60.76 [28 to 75] | 59.5 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 21 | 46
Weight in kilogram (kg) [Mean (Full Range); unit: kilograms] | 78.55 [57.5 to 144.9] | 78.76 [48.1 to 106.4] | 78.65 [48.1 to 144.9]
Length of hospital stay in days [Mean (Full Range); unit: Days] — Length of hospital stay. This is based the date of surgical procedure to the date of discharge from the hospital.
  Days | 3.88 [1 to 10] | 3.1 [0 to 6] | 3.5 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be the Percentage of Intraoperative Time the Participants Body Temperature is Above 36 Degrees Celcius.
Description: The total percent of intraoperative time (time in the operating room) that the body temperature of the participant is above 36 degrees celcius measured using an esophageal temperature probe.
Time Frame: 1 day
Measure: Mean (Full Range); unit: percent time
Arm/Group | Group 1: VitaHeat | Group 2: Bair Hugger
Number analyzed (Participants) | 25 | 21
percent time | 47.1 [0 to 100] | 72.0 [0 to 100]

2. Secondary Outcome: Post Operative Temperature on Admission to Post Operative Care Unit (PACU)
Description: Oral temperature in degrees celcius immediately after admission to the PACU after the planned surgical procedure has been completed.
Time Frame: Immediately after surgery
Population: 1 subject from the VITAheat group and 3 subjects from the Bair hugger group were excluded from analysis.
Measure: Mean (Full Range); unit: Degrees Celcius
Arm/Group | Group 1: VitaHeat | Group 2: Bair Hugger
Number analyzed (Participants) | 25 | 21
Degrees Celcius | 36.6 [35.0 to 37.3] | 36.8 [36.4 to 37.2]

ADVERSE EVENTS:
Time Frame: Up to 30 days after surgical procedure.
Arm/Group | Group 1: VitaHeat | Group 2: Bair Hugger
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/21
Other Adverse Events (participants affected / at risk) | 3/25 | 2/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VitaHeat (N=25) | Group 2: Bair Hugger (N=21)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) — Myocardial infarction during the planned surgical procedure.
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) — Cardiac arrest during the period of surgical start to the day of discharge.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VitaHeat (N=25) | Group 2: Bair Hugger (N=21)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 0 (0) — Urinary tract infection documented after surgical procedure to the time of discharge from the hospital.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Pneumonia reported during the time postsurgical to day of discharge from the hospital
Bladder injury (Renal and urinary disorders) | 0 (0) | 1 (1) — Bladder injury during the perioperative period.
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Deep vein thrombosis identified during the period of surgical date to the day of discharge,.
Device burn injury to skin (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Burn injury to skin related to the warming devices from surgical start time to end of surgery.

LIMITATIONS AND CAVEATS:
The limitation of the results presented is that we did not reach full enrollment as referenced in the protocol because the sponsor terminated the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT00913978/Prot_SAP_000.pdf